CLINICAL TRIAL: NCT06918704
Title: Behavioral Intervention Development Core - Working Memory Digital Intervention in Aging
Brief Title: BID WM Digital Intervention in Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-42925; P30AG086635 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Working Memory; Inhibitory Control; Mild Cognitive Impairment (MCI); Aging
Keywords: Cognitive Training; Working Memory; MCI; Inhibitory Control; Mild Cognitive Impairment; Aging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coherence Intervention (Active Comparator): Participants in this arm will engage with the Coherence Intervention.
  Interventions: Behavioral: Coherence
- Worder Intervention (Active Comparator): Participants in this arm will engage with the Worder intervention.
  Interventions: Behavioral: Worder

INTERVENTIONS:
Behavioral: Coherence — Coherence is a music-based rhythm training app.
  Arms: Coherence Intervention
Behavioral: Worder — Worder is a word search app.
  Arms: Worder Intervention

SUMMARY:
The goal of this clinical trial is to learn if engaging with an digital intervention may improve cognitive function. The main questions it aims to answer are:

1. Does engagement in with a digital intervention improve working memory?
2. Does engagement in with a digital intervention improve inhibitory control?

Researchers will compare two different digital interventions to assess whether they may be helpful in improving cognitive function.

Participants will conduct study activities remotely (e.g., at-home):

1. Baseline Assessment. Complete a series of cognitive assessments and surveys.
2. Intervention. Engage in a digital intervention for up to 8 weeks.
3. Post Intervention Assessment. Complete the same cognitive assessments and surveys as the Baseline Assessment.
4. Follow-Up Assessment. Six months after the intervention ends, participants will complete the same cognitive assessments and surveys as the Baseline Assessment.

DETAILED DESCRIPTION:
During the Baseline Assessment, participants will complete web-based cognitive assessments and surveys. The assessments will address various cognitive functions including working memory, long-term memory, inhibitory control, and sustained attention. Surveys will include a characterization of expectancy for the intervention, ratings of stress, and background health information. The Baseline Assessment will take up to 120 minutes and can be completed across more than one session.

During the Intervention, participants will be provided an iPad tablet to engage with the assigned intervention app. Participants will be randomly assigned to one of two intervention apps. Regardless of the assigned intervention, participants will engage with the app for 25-45 minutes of training per day, 5 days a week for up to 8 weeks for a total of 1000 minutes of training.

After the intervention, participants will complete a Post Intervention Assessment and 6 month later, a Follow-Up Assessment. Both of these assessment periods will consist of the same cognitive assessments and surveys as conducted during the Baseline Assessment.

Upon completion of all study activities, participants will be able to keep the iPad as a gift for their voluntary participation.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 12 years of education
* English fluency
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal vision
* Medically healthy older adults including those with below-average cognitive performance or mild cognitive impairment patients without dementia

Exclusion Criteria:

* Under the age of 60
* Clinical diagnosis of neurological or psychiatric disorder
* Visually or hearing impaired without correction to normal
* Clinical diagnosis of dementia or AD8 score of >3
* Regularly (one or more times per week) practicing an instrument within the last year
* 10 or more years of formal musical instrument training

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Working Memory | Immediately before the intervention, Immediately after the intervention, 6 months after the intervention
  Working memory performance will be assessed with a delayed match-to-sample task.

SECONDARY OUTCOMES:
Inhibitory Control | Immediately before the intervention, Immediately after the intervention, 6 months after the intervention
  Inhibitory control will be assessed with the Stroop task.
Inhibitory Control | Immediately before the intervention, Immediately after the intervention, 6 months after the intervention
  Inhibitory control performance will be assessed by distractors within a delayed match-to-sample task.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Zanto, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data to be shared includes demographic, cognitive assessments, survey, and behavioral outcomes.
Supporting Information: Study Protocol, ICF, Analytic Code